CLINICAL TRIAL: NCT03101657
Title: Evaluation of the Total Incapacity of Work (I.T.T.) in the Victims of Psychotraumatism Taken Care of in the Medico-judicial Unit of the CHU of Montpellier by Forensic Doctors and Psychologists
Brief Title: Evaluation of Total Disability (I.T.T.) in Victims of Psychotraumatism.
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0102
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-03

CONDITIONS: Psychotraumatism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The increase in psychological violence in our society, but also and above all the search for the best possible reparation for this violence, leads increasingly to questioning the evaluation of psychotraumatisms. In practice, there is no consensus as to the method of assessing psychological repercussions and determining ITI. This topic concerns any physician

DETAILED DESCRIPTION:
The increase in psychological violence in our society (psychological repercussions of physical violence, situations of harassment, psychotraumatism linked to the series of attacks suffered in France), but also and above all, the search for the best possible reparation for this violence The victims and the society), leads increasingly to question the evaluation of psychotraumatisms. In practice, there is no consensus as to the method of assessing psychological repercussions and determining ITI. This topic concerns any physician involved in the care of victims, whether he is a doctor in primary care or in specialized care.

ELIGIBILITY:
Inclusion criteria:

* Patients over 18 years of age taken in charge at the Médico-Judiciaire Unit of the CHU Montpellier following a physical and / or psychological traumatism. - - Starting up between 01.01.2016 and 31.12.2016.
* Patients who have undergone a double assessment (medical and psychological).

Exclusion criteria:

* Patients under the age of 18 years.
* Consultation within the framework of a takeover started before 01.01.2016.
* Absence of double medical and psychological evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients suffering from psychotraumatism.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Medico-psychological interviews | 1 day
  Study of standardized questionnaires resulting from medico-psychological interviews, the data of which will have been gathered during consultations as part of the care

CONTACTS AND LOCATIONS:
Overall Officials: thomas PERROT, Interne, Principal Investigator — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided
NC